CLINICAL TRIAL: NCT04030429
Title: Phase II Trial of Crizotinib in c-MET Mutation Metastatic/Recurrent/Persistent Endometrial Cancer
Brief Title: Crizotinib in c-MET Mutation Metastatic/Recurrent/Persistent Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patients were recruited during screen phase but fewer patients met criteria.
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Chi Mei Medical Hospital (Other); Kaohsiung Medical University (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-108-016
Record Dates: First submitted 2019-05-24; First posted 2019-07-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2022-04

CONDITIONS: Endometrial Cancer Recurrent
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Crizotinib arm (Experimental): Crizotinib 250 mg bid orally
  Interventions: Drug: Crizotinib 250 MG

INTERVENTIONS:
Drug: Crizotinib 250 MG — bid orally
  Other Names: Xalkori 250 MG

SUMMARY:
The majority of endometrial cancer patients with disease spread beyond the uterus will progress within 1 year. Platinum-based chemotherapy was used as the first-line treatment in metastatic or advanced endometrial cancer. There is no standard protocol for the second-line option when tumors persist or recur. In vitro and in vivo studies showed Crizotinib, an approved drug for the treatment of ALK-positive non-small cell lung cancer, demonstrated activities in endometrial cancer with c-MET kinase and Sema domain mutations. As a consequence, a phase 2 clinical trial to investigate the efficacy of Crizotinib in endometrial cancer patients with MET mutation is initiated.

DETAILED DESCRIPTION:
In this phase 2 study, the target population is patients with recurrent or persistent metastatic endometrial cancer. The mutation status of c-MET gene will be tested and only patients with c-MET mutation will be enrolled. After enrollment, Crizotinib 250 mg bid will be used orally. CT scan or MRI will be used to determine the response. Crizotinib will be continued till disease progression. Primary end is objective response rate. The secondary endpoints include progression-free survival, overall survival and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age no less than 20 years and no more than 75 years, at the time of acquisition of informed consent.
* Histological confirmed epithelial endometrial cancer
* Disease recurrent after curative therapy or adjuvant therapy including surgery, chemotherapy, radiotherapy or hormone therapy
* Metastatic/recurrent/persistent endometrial cancer
* Tumor tissue with high expression in immunohistochemistry stain (IHC) or somatic c-MET mutation
* Patients with symptomatic recurrent lesion or Image diagnosis (including ultrasound, Computed Tomography or Magnetic Resonance Imaging) recurrent status
* ECOG Performance status 0-2
* At least one distinct tumor, not previous irradiated, measurable lesion according to RECIST (version 1.1)
* Adequate organ function

Bone marrow:

Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L WBC ≥ 3.0 x 10^9/L Platelet count ≥ 100 x 10^9/L Hemoglobin ≥ 9 g/dL

Hepatic:

Total bilirubin level ≤ 1.0 x UNL AST and ALT ≤ 3.0 x UNL Renal: Creatinine level ≤ 1.5 mg/dL in men, ≤1.4 mg/dL in women; or Estimated CCr ≥ 60 mL/min (CCr is estimated by Cockcroft-Gault formula)

* Negative pregnancy test for women of childbearing potential only
* Patient willing to provide blood sample for research purposes
* Written informed consent

Exclusion Criteria:

* Presence or history of malignancy disease other than endometrial cancer that has been diagnosed with past five years
* Other anti-tumor agent such as systemic chemotherapy, hormone therapy or surgery within 2 weeks before the commencement of study treatment or radiotherapy within 4 weeks before the commencement of study
* Active uncontrolled infection
* Significant medical diseases, such as unstable angina, acute or recent myocardial infarction (<6 months before enrollment), COPD with frequent exacerbation, uncontrolled hypertension, ore cent CVA (<6 months before enrollment)
* Poor compliance
* Pregnant or breastfeeding women, where pregnancy is confirmed by a positive hCG laboratory test.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in best overall response rate | CT scan or MRI will be done at baseline and at the end of every 2 cycles (each cycle is 28 days) until the date of first documented progression or date of death from any cause, whichever came first, up to 104 weeks
  CT scan or MRI will be used to evaluate the response every 2 cycles according to the RECIST 1.1 criteria. The best overall response rate is the proportion of patients in whom a complete response (CR) or partial response (PR) was observed.

SECONDARY OUTCOMES:
Progression-free survival | CT scan or MRI will be done at baseline and at the end of every 2 cycles (each cycle is 28 days) until the date of first documented progression or date of death from any cause, whichever came first, up to 104 weeks
  CT scan or MRI will be used to evaluate the response according to RECIST 1.1 criteria. Progression-free survival is defined as the time from the time of treatment to disease progression or death from any cause.
Overall survival | Overall survival will be followed from the start of treatment to death from any cause, up to 104 weeks
  Overall survival is defined as defined as the time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Fu Hsu, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No